CLINICAL TRIAL: NCT01529996
Title: Comparison of the Efficacy Between Pulsed Dye Laser (PDL) and the Microsecond 1064-nm Nd:YAG Laser for Treatment of Diffuse Facial Redness: A Pilot, Prospective Randomized Trial.
Brief Title: Pulsed Dye Laser (PDL) vs. Microsecond 1064-nm Nd:YAG Laser for Treatment of Diffuse Facial Redness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU55489
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- YAG laser (Experimental)
  Interventions: Procedure: Pulse Dye Laser/YAG laser
- Pulse Dye Laer (Active Comparator)
  Interventions: Procedure: Pulse Dye Laser/YAG laser

INTERVENTIONS:
Procedure: Pulse Dye Laser/YAG laser — This study involves treatments with two types of lasers, Pulsed dye lasers (PDL) and the 1064 nm Nd: YAG. Both lasers are FDA approved to treat vascularities in the skin.

SUMMARY:
The primary objective of this study is to compare the efficacy of PDL and the 1064-nm Nd:YAG laser in the treatment of facial redness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients 18-55 years of age with erythematotelangiectatic rosacea (as verified by the the PI).
* Subjects who are willing to provide informed consent for participation in the study.

Exclusion Criteria:

* Pregnant or lactating individuals
* Subjects who are unable to understand the protocol or to give informed consent.
* Subjects who have a known history of photosensitive conditions (e.g. Systemic lupus, polymorphous light eruption)
* Subjects who have facial telangiectasia of diameter greater than 2 mm.
* Subject who have significant (as determined by the PI) acute inflammatory papules, pustules, and vesicle involving the central face.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Rating on global improvement scale | four months
  Non-treating dermatologists will rate each side of the face using a global improvement scale to evaluate the effectiveness of the two treatments.
Spectrophotometer measurement | four months
  Spectrophotometer measurement as the percent resolution on each follow up visit compared to baseline visit

SECONDARY OUTCOMES:
Patient satisfaction | four months
  Patients will record satisfaction on the questionnaires provided
Recorded discomfort | four months
  Subjects will record discomfort using a 10-point scale
Adverse events | four months
  Any adverse events will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States